CLINICAL TRIAL: NCT01111201
Title: Pilot Survey to Assess International Travel Patterns and Risk Behaviour of Breast Cancer, Lymphoma Patients and Bone Marrow Transplant Recipients at Memorial Sloan-Kettering Cancer Center
Brief Title: International Travel Patterns and Risk Behaviour of Breast Cancer, Lymphoma Patients and Bone Marrow Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-045
Record Dates: First submitted 2010-04-22; First posted 2010-04-27 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer; Lymphoma
Keywords: Autologous Bone Marrow Transplant; Breast; Lymphoma; International travel; questionnaire; Hematopoietic Stem Cell Transplant (HSCT) recipients
MeSH Terms: conditions — Breast Neoplasms; Lymphoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- questionnaires: There will be four versions of the questionnaire, each slightly modified to be more specific toward the treatment paradigms in the respective target patient population (Breast Cancer/ Lymphoma/Autologous Bone Marrow Transplant/ Allogeneic Bone Marrow Transplant). All questionnaire versions will consist of seven sections.
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — The intervention is a self-administered anonymous questionnaire that is voluntarily completed by the patient. Questions in Section One will cover general information about the patient including gender, age, race, country of birth, current zip code of residence, and level of education. Questions in Section Two will cover information regarding the cancer (breast/lymphoma) or transplant (allogeneic/ autologous). Questions in Section Three will cover travel history including the frequency of travel outside the United States and Canada in the last 5 years. Questions in Sections Four through Seven will obtain information about their last trip outside the United States and Canada.

SUMMARY:
This study also aims to raise awareness among both patients and health-care providers about the importance of pre-travel health consultation and preventive interventions prior to international travel.

Through appropriate health counseling, cancer patients will have less risk of having travel -related health complications and thus have a better quality of life and overall improved sense of wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Hematopoietic Stem Cell Transplant (HSCT) recipients
* Age >18 years
* Status post bone marrow transplant within last five years Breast Cancer patients: Criteria 1 and Criteria 2 and/or 3
* Female age >18 years and current or past history of breast cancer
* Received systemic chemotherapy in the last five years
* Metastatic breast cancer disease (stage IV) Lymphoma: Criteria 1 and Criteria 2 and/or 3
* Age >18 years and current or past history of lymphoma
* Received systemic chemotherapy within 5 years
* Had active disease at any time within the last 5 years

Exclusion Criteria:

* Patients age< 18 years
* Breast cancer and lymphoma patients in clinical remission in the past 5 years
* Patients unable to fill the questionnaire due to language barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The goal accrual is 50 patients from each of the following oncology services:
  Breast, Lymphoma, Autologous Stem Cell Transplant, and Allogeneic Stem Cell Transplant.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To determine the frequency of international travel of the targeted patients in the last 5 years. | once at the time of the clinic visit

SECONDARY OUTCOMES:
To determine if any of the international travel was during a high-risk specific period when the immune status of the target population was compromised. | once at the time of the clinic visit
To profile the target population who traveled internationally with respect to their demographic and cancer/transplant-related characteristics. | once at the time of the clinic visit
To obtain detailed information about their last international trip including | once at the time of the clinic visit
To assess the adequacy of the questionnaire instructions | once at the time of the clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Monika Shah, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org